CLINICAL TRIAL: NCT03062124
Title: Single-operator Peroral Pancreatoscopy in Preoperative Diagnostics of Presumed Main Duct Intraductal Papillary Mucinous Neoplasms: Efficacy and Novel Insights on Complications
Brief Title: SpyGlass in Preoperative Diagnostics of Presumed Main Duct IPMNs: Efficacy and Novel Insights on Complications
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leena Kylanpaa, MD, PhD, Helsinki University Central Hospital
Other Study IDs: IPMN SpyGlass
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Intraductal Papillary Mucinous Neoplasm
Keywords: SpyGlass; Pancreatoscopy; Single-operator pancreatoscopy; post-ERCP pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — * Tissue biopsies collected from suspected IPMN (Intraductal Papillary Mucinous Neoplasm) lesions
  * Flushing fluid from pancreatic duct
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: SpyGlass pancreatoscopy — During the SpyGlass pancreatoscopy procedure visually guided biopsies and flushing liquid are collected from the pancreatic duct

SUMMARY:
Distinguishing intraductal papillary mucinous neoplasms (IPMNs) from other pancreatic cystic lesions is essential as IPMNs bear risk of becoming malignant. Differentiating the main pancreatic duct involving IPMNs (MD-IPMNs) with imaging can be difficult. Single-operator peroral pancreatoscopy (SOPP) has shown to be a promising method offering additional information on suspected lesions in the main pancreatic duct (MD). We aimed to establish the role of SOPP in preoperative diagnostics of presumed MD-IPMNs. A secondary objective was to identify factors that contribute to SOPP-related complications.

DETAILED DESCRIPTION:
In this multicenter, partly prospective, but mostly retrospective cohort study, 101 SOPPs were performed due to presumed MD-IPMNs in three centers. As a key outcome, the rate of how often visual appearance of MD, and/or MD flushing liquid samples and biopsies taken during SOPP affected further clinical care, was determined. Secondly, post-SOPP complications according to Cotton consensus criteria, diameter of MD, use of prophylactic nonsteroidal anti-inflammatory drugs (NSAIDs) and pancreatic stents, duration of SOPP and timing of pancreatic sphincterotomy (PS) were documented.

ELIGIBILITY:
Inclusion Criteria:

* Medical imaging showing suspision of IPMN,.
* Medical imaging showing dilatation of the pancreatic duct

Exclusion Criteria:

- Malignancy confirmed by previous examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter study, patients from Helsinki University Hospital, Skåne University Hospital and Karolinska University Hospital. All patients underwent single-operator peroral pancreatoscopy due to presumed main duct IPMNs
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Histologic diagnosis given by the collected samples | 1 year
  Pathologists report
Influence in decision-making concerning the patients clinical management | 1 year
  Multidisplinary meeting decision after SpyGlass

SECONDARY OUTCOMES:
Post procedural complications emerged after SpyGlass pancreatoscopy | 1 year
  According to Cotton criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sini M Vehviläinen, MD, Study Chair — Helsinki University Central Hospital; Hanna Seppänen, MD, PhD, Study Chair — Helsinki University Central Hospital; Marianne Udd, MD, PhD, Study Chair — Helsinki University Central Hospital; Outi Lindström, MD, PhD, Study Chair — Helsinki University Central Hospital; Leena Kylänpää, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Urban Arnelo, Study Chair — Karolinska University Hospital; Niklas Fagerström, Study Chair — Karolinska University Hospital; Roberto Valente, Study Chair — Karolinska University Hospital; Harri Mustonen, Study Chair — Helsinki University Central Hospital; Fredrik Swahn, Study Chair — Skane University Hospital
Locations (3):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnelo U, Siiki A, Swahn F, Segersvard R, Enochsson L, del Chiaro M, Lundell L, Verbeke CS, Lohr JM. Single-operator pancreatoscopy is helpful in the evaluation of suspected intraductal papillary mucinous neoplasms (IPMN). Pancreatology. 2014 Nov-Dec;14(6):510-4. doi: 10.1016/j.pan.2014.08.007. Epub 2014 Sep 27. PMID 25287157
- [Background] Tanaka M, Fernandez-del Castillo C, Adsay V, Chari S, Falconi M, Jang JY, Kimura W, Levy P, Pitman MB, Schmidt CM, Shimizu M, Wolfgang CL, Yamaguchi K, Yamao K; International Association of Pancreatology. International consensus guidelines 2012 for the management of IPMN and MCN of the pancreas. Pancreatology. 2012 May-Jun;12(3):183-97. doi: 10.1016/j.pan.2012.04.004. Epub 2012 Apr 16. PMID 22687371